CLINICAL TRIAL: NCT04642508
Title: The PreQ-20 TRIAL, a Prospective Cohort Study of the Oncologic Safety, Quality of Life and Cosmetic Outcomes of Patients Undergoing Prepectoral Breast Reconstruction
Brief Title: The PreQ-20 TRIAL, a Prospective Cohort Study of Patients Undergoing Prepectoral Breast Reconstruction
Acronym: PreQ-20
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Benigno Acea, Breast Surgeon, University Hospital A Coruña
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/295
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Quality of Life; Surgery--Complications
Keywords: Prepectoral Reconstruction; Sparing Mastectomy; Risk reducing mastectomy; Breast Q
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prepectoral Reconstruction (Other): Women with breast cancer or with high risk for breast cancer in whom a sparing mastectomy and prepectoral reconstruction was performed
  Interventions: Procedure: Prepectoral reconstruction

INTERVENTIONS:
Procedure: Prepectoral reconstruction — Immediate prepectoral breast reconstruction in women requiring a mastectomy

SUMMARY:
The investigators conducted a prospective cohort study to assess the safety, quality of life and cosmetic sequelae of prepectoral breast reconstruction in women with breast cancer and high risk. The study's main objective is to assess the safety of prepectoral breast reconstruction in terms of postsurgical complications and the feasibility of reconstruction (loss of implants). The secondary objectives are to evaluate oncologic safety (local relapses, residual glandular tissue) and to identify factors related to quality of life and cosmetic sequelae. The evaluation of residual tissue will be conducted by magnetic resonance imaging 12 to 18 months after the surgery, and the quality-of-life assessment will be performed using the BreastQ questionnaire. An initial patient evaluation will be conducted 12-18 months after the surgery, and a second evaluation will be performed at 5 years. The estimated sample size is 81 patients.

DETAILED DESCRIPTION:
1. Mastectomy technique. The breast removal will be performed using a mastectomy adapted to the breast and optimizing the preservation of the breast's original elements (inframammary fold, skin envelope, fat transitions, nipple-areolar complex) according to each patient's anatomical and oncologic possibilities.
2. Reconstruction technique. The reconstruction will be performed by placing a silicone implant coated with polyurethane foam in the prepectoral position.
3. Preoperative assessment. All patients will be assessed by a surgeon of the breast unit. The decision for the mastectomy will be made in consensus with the multidisciplinary committee. Before the surgery, the patients will undergo a mammography and magnetic resonance imaging to confirm the tumor size and rule out multifocality/multicentricity, as well as an evaluation of the distribution of glandular tissue and transitions between the breast and chest wall.
4. Breast magnetic resonance imaging. This study will employ the first magnetic resonance imaging during the postoperative period (between 12 and 18 months) to assess the residual glandular tissue following the mastectomy.
5. BreastQ questionnaire. The BreastQ questionnaire is aimed at evaluating patient-reported satisfaction and quality of life through the use of breast reconstruction modules. The preoperative format, which is delivered to patients before the surgery, and the postoperative format, which is delivered to them 12-18 months after the surgery. Likewise, we will conduct a second postoperative assessment at 5 years of the surgery.

d. Images. The evaluation of the cosmetic sequelae requires taking photographs of the patient's chest (from the suprasternal notch to navel). Photographs will be taken prior to the surgery (frontal, right and left lateral), then again at 12-18 months and finally at 5 years of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* We will include all women operated on in the Breast Unit through skin sparing mastectomy/Nipple skin sparing mastectomy (unilateral or bilateral) and immediate reconstruction with prepectoral implantation.

The study population will include 2 patient groups:

1. Women with breast carcinoma. This group consists of patients with a histological diagnosis of in situ or infiltrating breast carcinoma, either primary or metachronic, which requires mastectomy as the surgical treatment.
2. Women at high risk for breast cancer. This group consists of women evaluated at a high-risk consultation and whose reducing risk mastectomy has been approved by the tumor committee of the Breast Unit of University Hospital Complex of A Coruna. For this procedure, the patients should meet at least one of the following criteria:

   * Hereditary breast and ovarian cancer syndrome, either by demonstrated genetic mutation or through their family history.
   * Histological diagnosis of high-risk lesions (atypical hyperplasia, ductal carcinoma in situ, lobular carcinoma in situ) associated with family history.
   * High-risk criteria (genetic, histological, family) during the breast cancer follow-up.

Exclusion Criteria:

* Inability to undergo magnetic resonance imaging during the diagnosis and follow-up.
* Inability to fill out the BREAST-Q questionnaire.
* Unwillingness by the patient to participate in the study.
* Breast sarcomas.
* Benign breast tumors.
* Prepectoral breast reconstruction using expanders.
* Prepectoral reconstruction with mesh

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of implant loss (Feasibility of recosntruction) | First year after surgery
  To evaluate the feasibility of prepectoral reconstruction in terms of implant loss the first year after surgery, also during oncological treatment (example: chemotherapy) (Unit of mesure: number of implant loss)
Incidence of surgical complications - reoperations (Safety) | 3 months after surgery
  To determine the global incidence of surgical complications, as well as the causes of complications in terms of: postoperative bleeding, skin necrosis, necrosis of the nipple areola complex, seroma and infection

SECONDARY OUTCOMES:
Incidence of residual glandular tissue (Safety) | 1 year after surgery
  To evaluate the safety of sparing mastectomy through the identification of residual glandular tissue through a magnetic resonance one year after surgery
Incidence of breast cancer relapse (oncological safety) | yearly, up to 5 years. From surgery date until the date of documented realapse
  To evaluate the safety of sparing mastectomy through the identification relapses in the same breast during the follow up
Incidence of new breast cancer (safety of risk reducing mastectomy) | yearly, up to 5 years. From surgery date until the date of documented new breast cancer
  To evaluate the safety of risk reducing sparing mastectomy in high risk for breast cancer patientes through the identification of new breast cancer
Quality of life and satisfaction after a mastectomy with prepectoral reconstruction, using the BreastQ questionnaire | 1 year and 5 year after surgery
  To assess satisfaction and quality of life after prepectoral reconstruction in women with breast cancer and those with high risk through breastQ questionnaire To identify factors related to satisfaction and quality of life after prepectoral reconstruction (e.g. marital status, psychological illnesse)
Incidenca of cosmetic sequelae | yearly, up to 5 years. From surgery date until the date of first documented cosmetis sequelae
  To evaluate the cosmetic sequelae after prepectoral reconstruction in women with breast cancer and with high risk and Identify factors related to the cosmetic sequelae after prepectoral reconstruction. The investigators will employ the Clough classification, where type I sequelae identified the patients with breast asymmetry but no deformity, type II sequelae were defined by the presence of a deformity that could be corrected using a breast-conserving procedure, and type III sequelae identified those women whose breast showed a deformity or painful fibrosis that could only be solved through mastectomy. To determine the sequelae, the criteria of the breast surgeon will be used, documented through photos.

CONTACTS AND LOCATIONS:
Overall Officials: Benigno Acea Nebril, PhD., Principal Investigator — University Hospital A Coruña
Locations (1):
- Hospital Abente y Lago, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acea-Nebril B, Garcia-Novoa A, Garcia Jimenez L. The PreQ-20 TRIAL: A prospective cohort study of the oncologic safety, quality of life and cosmetic outcomes of patients undergoing prepectoral breast reconstruction. PLoS One. 2022 Jul 14;17(7):e0269426. doi: 10.1371/journal.pone.0269426. eCollection 2022. PMID 35834508